CLINICAL TRIAL: NCT00620789
Title: Behavioral Insomnia Therapy For Those With Insomnia and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Colleen Carney, PhD, Department of Psychology, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00003416; 1R01MH076856-01A2 (NIH)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Insomnia; Major Depressive Disorder
Keywords: Insomnia; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Cognitive-Behavior Therapy for insomnia (CBT-I) + Antidepressant medication
  Interventions: Drug: Escitalopram + CBT-I
- 2 (Placebo Comparator): Cognitive Behavior Therapy for Insomnia (CBT-I) + placebo medication
  Interventions: Behavioral: CBT-I plus placebo antidepressant medication
- 3 (Sham Comparator): Antidepressant medication + Sleep Hygiene Control (SH)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram + CBT-I — * Escitalopram, 10 mg daily for the duration of the study (6 months)
  * CBT-I, four biweekly sessions during eight week Treatment phase.
  Other Names: Escitalopram,Lexipro; CBT-I, Cognitive Behavioral Therapy-Insomnia
  Arms: 1
Behavioral: CBT-I plus placebo antidepressant medication — * CBT-I, 4 biweekly sessions, eight week Treatment phase.
  * Placebo,daily for duration of study(6 months).
  Other Names: CBT-I, Cognitive Behavioral Therapy Insomnia
  Arms: 2
Drug: Escitalopram — * Escitalopram, 10 mg daily for the duration of the study (6 months)
  * SH, four biweekly sessions during eight week Treatment phase
  Other Names: Escitalopram, Lexipro; SH,Sleep Hygiene
  Arms: 3

SUMMARY:
This study is a randomized clinical trial to test the efficacy of Cognitive-Behavioral Insomnia Therapy when used in isolation or in combination with antidepressant medication (escitalopram) among patients with Major depressive disorder and insomnia.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a highly prevalent and debilitating condition that reduces quality of life, increases health care utilization, markedly impairs social/occupational functioning, and enhances suicide risk for countless individuals worldwide. A substantial proportion of MDD patients present with comorbid insomnia that significantly complicates their clinical management. For many such patients, insomnia represents a longstanding and problematic condition that predates the onset of MDD, adds to their suicide risk, dampens their response to traditional depression treatment, and enhances the likelihood for MDD relapse. Moreover, many patients who show remission of depressive symptoms with traditional therapies (e.g., antidepressant medications, cognitive therapy) suffer from residual insomnia that increases their chances for eventual relapse. Despite the deleterious effects insomnia may have on MDD patients, there has been surprisingly little research to test effective insomnia management strategies among this patient group. Some reports suggest that depression treatments may benefit from adding a hypnotic medication to traditional depression therapy, but this approach has it limits since sleep improvements achieved with hypnotics do not endure after hypnotic discontinuation. Cognitive-Behavioral Insomnia Therapy (CBT-I) represents a promising alternative treatment for MDD since it is highly effective and produces sleep improvements that persist well beyond the discontinuation of acute therapy. Unfortunately CBT-I has yet to be tested among MDD patients with comorbid insomnia. In the current project, we will conduct a randomized clinical trial to test the efficacy of CBT-I when used in isolation or in combination with antidepressant medication (escitalopram) among MDD patients with comorbid insomnia. A sample of 201 patients with MDD and comorbid insomnia will be randomized to treatments consisting of the combination of antidepressant medication plus CBT-I, antidepressant medication plus placebo behavioral insomnia therapy, or CBT-I plus a placebo medication. Objective (polysomnography, actigraph) and subjective (sleep diary, questionnaires) sleep measures, as well as depression and quality of life measures will be obtained before therapy, after an 8-week treatment phase, and at 6-months follow-up. Results of this trial will provide important new information about the short and long-term management of those highly challenging and difficult to treat patients with insomnia comorbid to MDD.

Hypothesis I asserts that the combined CBT-I+AD therapy will produce significantly greater pre-to-post therapy improvements in sleep continuity measures than will the 2 mono-therapy conditions. The primary outcomes for these hypotheses are subjective (sleep diary) measures of TWT and SE. These sleep measures are recorded daily for 2-week periods at baseline, post-treatment, and the 6-month follow-up. The daily measures will be averaged over each 2-week period. As a result, patients will have three repeated outcomes for each of the two sleep measures: one representing the average at baseline, one for the average at post-treatment, and one for the average at 6-months. Sleep diary estimates of TWT and SE from pre to post treatment will serve as the primary measures to test this hypothesis. Our secondary outcome measures include diary estimates of total sleep time (TST), as well as objective measures of TWT, SE, & TST taken from pre-and post-treatment PSG and actigraphic monitoring We will use a 3 (treatment groups) x 2 (Baseline vs. post-treatment) Analysis of Variance (ANOVA) model to compare the performance of our treatment conditions across the primary and secondary outcomes. Treatment comparisons of CBT-I + AD vs. each of the other 2 treatments will be made. Alpha for the 2 primary outcomes is fixed at 0.025 (= 0.05/2). Further analyses will adjust for pre-treatment stratification variables and other covariates. The investigators will, in particular, be mindful of the treatment adherence and credibility data we collect and use these measures as covariates if the investigators find differential adherence or credibility rates across treatment conditions. In addition, the investigators will explore the effect of changes in medication on the observed changes in our outcome measures by considering medication usage data derived from the MQS106.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-64 years old
* insomnia complaint of at least one month duration that meets the Research Diagnostic Criteria for Insomnia
* meet DSM-IV criteria for a Major Depressive Episode (without psychotic features) as verified by the mood module of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID

Exclusion Criteria:

* need immediate psychiatric (e.g., imminently suicidal patients) or medical care (e.g., patients with acute cardiac symptoms), or have attempted suicide in the past 6 months
* have a sleep-disruptive comorbid medical condition (e.g., moderate to severe rheumatoid arthritis
* are pregnant, trying to get pregnant, or not currently practicing adequate birth control methods
* score < 27 on the Mini-Mental Status Exam
* meet DSM-IV criteria for Obsessive-Compulsive disorder, Generalized Anxiety Disorder, Post-Traumatic Stress Disorder, Acute Stress Disorder, Panic Disorder, Bipolar Disorder, Schizophrenia or any other psychotic disorders on the basis of a SCID interview
* meet DSM-IV criteria for Antisocial Personality Disorder or Borderline Personality Disorder on the basis of a SCID II interview schedule
* report frequent travel across time zones or work rotating or night shifts
* meet criteria for sleep apnea, restless legs syndrome or Circadian Rhythm Sleep Disorder on the basis of the Duke Structured Interview of Sleep Disorders (DSISD)
* have an apnea-hypopnea index > 15 or periodic limb movement-related arousal index > 15 per hour of sleep during a screening laboratory polysomnogram
* have a history of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence in the 6 months prior to screening or have a positive urine drug or alcohol test at the time of screening
* report having taken the study drug (escitalopram) for 28 days or more and then discontinuing the medication due to side effects or adverse event
* have a disorder characterized by altered metabolism, a seizure disorder, severe renal impairment, a history of upper gastrointestinal bleed disorder, or a history of a condition that could interfere with the absorption, distribution, metabolism, or excretion of escitalopram
* participated in any other investigational drug study within 30 days prior to screening or become enrolled in another such study during the time they are enrolled in the current project
* use of any drugs known or suspected to affect hepatic or renal clearance within 30 days prior to screening for the current project
* are taking any medications that interact with escitalopram (e.g., Cimetidine, Lithium, Sumatriptan, Carbamazepine, or Ketoconazole) and are not willing to both taper off such medications during a time period equal to more than five half lives before entering the study and abstain from such medications throughout the study
* are unwilling or unable to abstain from non-study prescription medications for sleep (e.g., sedative hypnotics) or depression during their time in the study
* are known to be seropositive for Human Immunodeficiency Virus (HIV).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 477 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Mean two-week sleep log estimate of post-treatment sleep continuity | An average of two-weeks post-treatment
  Mean two-week post-treatment sleep log sleep continuity

SECONDARY OUTCOMES:
Mean two-night polysomnographic post-treatment sleep continuity | An average of two-weeks post-treatment
  Mean two-night polysomnographic post-treatment sleep continuity

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Carney, PhD, Principal Investigator — Licensed, North Carolina Psychology Board, Ontario Psychological Association, Association for Behavioral and Cognative Therapies, ABCT Insomnia and other Sleep Disorders Special Interest Group, Sleep Research Society, American Academy of Sleep Medicine
Locations (1):
- Ryerson University, Toronto, Ontario, Canada